CLINICAL TRIAL: NCT04616872
Title: Treatment of Patients With Coronary and Aortic Atherosclerotic Disease With Methotrexate-associated to LDL Like Nanoparticles. A Randomized, Double-blind, Placebo-control Trial
Brief Title: Treatment of Patients With Atherosclerotic Disease With Methotrexate-associated to LDL Like Nanoparticles
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Raul Cavalcante Maranhão, MD; PHD. Director Lipid Metabolism Laboratory, Heart Institute, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4786/19/005
Record Dates: First submitted 2020-10-24; First posted 2020-11-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Inflammation
Keywords: Atherosclerosis; coronary artery disease; inflammation; methotrexate; nanoparticles; nanotechnology; drug delivery system
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-control Trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate-LDE (Experimental): Methotrexate carried by a lipid nanoparticle (MTX-LDE)
  Interventions: Drug: Methotrexate-LDE
- Placebo-LDE (Placebo Comparator): Lipid nanoparticle (LDE)
  Interventions: Drug: Placebo-LDE

INTERVENTIONS:
Drug: Methotrexate-LDE — MTX-LDE 40mg/m2 (250mL total volume) IV and Folic acid 5mg by mouth (the day after MTX-LDE) weekly for 12 weeks
  Arms: Methotrexate-LDE
Drug: Placebo-LDE — Placebo-LDE (250mL total volume) IV and Folic acid 5mg by mouth (the day after Placebo-LDE) weekly for 12 weeks
  Arms: Placebo-LDE

SUMMARY:
The investigators propose a prospective, randomized, double-blind, placebo-controlled study. The purpose of the study is to evaluate the safety and efficacy of an anti-inflammatory agent methotrexate in a cholesterol-rich non-protein nanoparticle (MTX-LDE) in patients with stable coronary disease.

Patients with multi-vessels stable coronary disease will be randomized to receive MTX-LDE IV or placebo-LDE IV each 7 days for 12 weeks. The primary and main secondary endpoints will be analyzed by coronary and aortic CT angiography, that will be performed before the first treatment cycle, four weeks after the last drug infusion and 12 months after randomization. Patients will undergo clinical and laboratory safety evaluations before each treatment cycle, four weeks after the last cycle and 12 months after randomization.

An algorithm for drug suspension based on clinical and laboratory finding will be followed.

DETAILED DESCRIPTION:
Atherosclerosis is a life-threatening condition, as long as cardiovascular disease is responsible for one-third of all global mortality.

Inflammation is extremely important in atherosclerosis pathophysiology. The use of inflammatory biomarkers to predict risk, monitor treatments and guide therapy, has shown substantial potential for clinical applicability. Many studies in primary and secondary prevention of cardiovascular disease showed that individuals with lower high sensitive C-reactive protein (hsCRP) have better clinical outcomes than those with higher levels.

The potential benefit of anti-inflammatory therapy in atherosclerosis has been previously demonstrated in studies in patients with chronic inflammatory diseases (rheumatoid arthritis, psoriasis). The use of methotrexate has been associated with a reduction in cardiovascular events in these patients.

In this setting, the use of non-invasive treatments to reduce lesion size and inflammation is essential for the prevention of sub-sequent cardiovascular events.

The systemic use of methotrexate at high doses for the treatment of atherosclerotic cardiovascular diseases is unlikely due to their significant, often life-threatening toxicity. Nonetheless, the toxicity of such agents can be strongly diminished by the use of optimized drug-delivery systems. In a pioneer study performed on patients with acute leukemia, was reported the potential of a cholesterol-rich non-protein nanoparticle (LDE) as a drug targeting agent. LDE particles have lipid compositions and structures that resemble low-density lipoprotein (LDL) and can be injected directly into the bloodstream. When LDE particles come into contact with plasma, the particles acquire exchangeable apolipoproteins from native lipoproteins, such as apolipoprotein (apo) E, which binds the particles to LDL receptors. In neoplastic cells, lipoprotein receptors are overexpressed, such that uptake of native LDL and of LDE particles is increased relative to that in normal tissues. In aortas of cholesterol-fed rabbits the uptake of LDE particles is increased in comparison to normal aortas and in rabbit-grafted hearts take up the nanoemulsion at amounts fourfold greater than native hearts.

LDE-methotrexate treatment of rabbits induced to exhibit atherosclerosis via high cholesterol intake resulted in a 65% reduction in lesion size.

The aim of this study is to investigate whether patients with aortic and coronary atherosclerotic disease showed good tolerability to LDE-methotrexate treatment and whether this formulation could achieve reduction in plaque volume and characteristics by coronary and aortic CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* Multi-vessels coronary artery disease diagnosis by coronary CT or invasive angiography
* Aortic atherosclerosis diagnosis by multidetector computed tomography (MDCT) angiography.
* High-sensitivity C reactive protein (hs-CRP) levels > 2mg/L
* Signing the study informed consent.

Exclusion Criteria:

* History of Acute myocardial infarction in the last 30 days
* Heart failure with ejection fraction <40%
* Estimated glomerular filtration rate < 40 mL/min/1.73 m2.
* Prior history of chronic infectious disease, including tuberculosis, severe fungal disease, or known HIV positive.
* Chronic hepatitis B or C infection.
* Prior history of nonbasal cell malignancy or myeloproliferative or lymphoproliferative disease within the past 5 years.
* White blood cell count <4000/mm3, hematocrit <32%, or platelet count <75000/mm3.
* Alanine aminotransferase levels (ALT) greater than 3-fold the upper limit of normal.
* History of actual alcohol abuse or unwillingness to limit alcohol consumption to < 4 drinks per week.
* Pregnancy or breastfeeding.
* Women of child bearing potential, even if currently using contraception.
* Men who plan to father children during the study period or who are unwilling to use contraception.
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers.
* Known chronic pericardial effusion, pleural effusion, or ascites.
* Angina pectoris Canadian Cardiovascular Society (CCS) III-IV
* New York Heart Association class III-IV congestive heart failure.
* Contraindication for the use of iodinated contrast
* Life expectancy of < 1 years.
* Acute or Chronic aortic dissection
* Interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis.
* Current indication for methotrexate therapy.
* Patient with a history of an allergic reaction or significant sensitivity to methotrexate.
* Requirement for use of drugs that alter folate metabolism (trimethoprim/sulfamethoxazole) or reduce tubular excretion (probenecid) or known allergies to antibiotics making avoidance of trimethoprim impossible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-10-12 (Estimated); Study Completion 2023-10-12 (Estimated)

PRIMARY OUTCOMES:
Low Attenuation Plaque Volume (LAPV) coronary | Baseline and change from baseline to 4 months.
  Compare Low attenuation Plaque Volume( LAPV) measured by coronary CT angiography between groups.
Low Attenuation Plaque Volume (LAPV) coronary | Baseline and change from baseline to 12 months
  Compare Low attenuation Plaque Volume( LAPV) measured by coronary CT angiography between groups.
Low Attenuation Plaque Volume (LAPV) aortic | Baseline and change from baseline to 4 months
  Compare Low attenuation Plaque Volume( LAPV) measured by aortic CT angiography between groups.
Low Attenuation Plaque Volume (LAPV) aortic | Baseline and change from baseline to 12 months
  Compare Low attenuation Plaque Volume( LAPV) measured by aortic CT angiography between groups.

SECONDARY OUTCOMES:
Noncalcified plaque volume (NCPV) | Baseline and change from baseline to 4 months
  Compare Noncalcified plaque volume (NCPV) measured by coronary CT angiography between groups.
Dense calcified plaque volume (DCPV) | Baseline and change from baseline to 12 months
  Compare Dense calcified plaque volume (DCPV) measured by coronary CT angiography between groups.
Total lumen value (TLV) | Baseline and change from baseline, 4 months and 12 months
  Compare Total lumen value (TLV) measured by coronary CT angiography between groups.
Remodeling index (RI) | Baseline and change from baseline, 4 months and 12 months
  Compare Remodeling index (RI) measured by coronary CT angiography between groups.
Perivascular fat attenuation index (FAI) | Baseline and change from baseline, 4 months and 12 months
  Compare Perivascular fat attenuation index (FAI) measured by coronary CT angiography between groups.
Total atheroma volume (TAV) | Baseline and change from baseline, 4 months and 12 months
  Compare Total atheroma volume (TAV) measured by coronary CT angiography between groups.
Total atheroma volume (TAV) aortic | Baseline and change from baseline, 4 months and 12 months
  Compare Total atheroma volume (TAV) measured by aortic CT angiography between groups.
Clinical significant symptoms | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare the incidence of clinical significant symptoms (new and persistent stomatitis, vomiting, diarrhea, unexplained cough with fever, shortness of breath, alopecia, neurotoxicity, myalgia, arthralgias, bradycardia, hypotension, local pain) reported in each visit between groups.
Other adverse events | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare the incidence of other adverse events (not expected) reported in each visit between groups.

OTHER OUTCOMES:
Red blood cell count | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare hemoglobin and hematocrits levels between groups.
White blood cell count | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare leucocyte and neutrophil levels between groups.
Platelet count | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare Platelet levels between groups.
Alanine aminotransferase (ALT) | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare Alanine aminotransferase (ALT) levels between groups.
Aspartate aminotransferase (AST) | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare Aspartate aminotransferase (AST) levels between groups.
Creatinine | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare Creatinine levels between groups.
Urea | 1; 2; 3; 4; 5; 6; 7; 8; 9; 10; 11; 12; 16 and 52 weeks after randomization
  Compare Urea levels between groups.
Inflammatory biomarkers | Baseline and change from baseline, 4 months and 12 months
  Compare High-sensitivity C reactive protein (hs-CRP); Interleukin 6 (IL-6); Interleukin 1b (IL-1b); Interleukin 10 (IL-10); Interleukin 8 (IL-8); Interleukin 17 (IL-17); Tumor necrosis factor-alpha (TNF-a); Interferon gamma (IFN-y) levels between groups.
Cholesterol | Baseline and change from baseline, 4 months and 12 months
  Compare Total Cholesterol; High-density lipoprotein cholesterol (HDL) ; Low-density lipoprotein cholesterol (LDL); Triglyceride levels between groups.
Cholesterol efflux | Baseline and change from baseline, 4 months and 12 months
  Compare Cholesterol efflux between groups.
Creatine phosphokinase (CPK) | Baseline and change from baseline, 4 months and 12 months
  Compare Creatine phosphokinase (CPK) levels between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Heart Institute (InCor) - University of São Paulo Medical School, São Paulo, Brazil, São Paulo, São Paulo
  - Institute Prevent Senior, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Maranhao RC, Vital CG, Tavoni TM, Graziani SR. Clinical experience with drug delivery systems as tools to decrease the toxicity of anticancer chemotherapeutic agents. Expert Opin Drug Deliv. 2017 Oct;14(10):1217-1226. doi: 10.1080/17425247.2017.1276560. Epub 2017 Jan 1. PMID 28042707
- [Background] Bulgarelli A, Leite AC Jr, Dias AA, Maranhao RC. Anti-atherogenic effects of methotrexate carried by a lipid nanoemulsion that binds to LDL receptors in cholesterol-fed rabbits. Cardiovasc Drugs Ther. 2013 Dec;27(6):531-9. doi: 10.1007/s10557-013-6488-3. PMID 24065615
- [Background] Shapiro MD, Fazio S. From Lipids to Inflammation: New Approaches to Reducing Atherosclerotic Risk. Circ Res. 2016 Feb 19;118(4):732-49. doi: 10.1161/CIRCRESAHA.115.306471. PMID 26892970
- [Background] van Diepen JA, Berbee JF, Havekes LM, Rensen PC. Interactions between inflammation and lipid metabolism: relevance for efficacy of anti-inflammatory drugs in the treatment of atherosclerosis. Atherosclerosis. 2013 Jun;228(2):306-15. doi: 10.1016/j.atherosclerosis.2013.02.028. Epub 2013 Mar 1. PMID 23518178
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Ridker PM. Residual inflammatory risk: addressing the obverse side of the atherosclerosis prevention coin. Eur Heart J. 2016 Jun 7;37(22):1720-2. doi: 10.1093/eurheartj/ehw024. Epub 2016 Feb 22. No abstract available. PMID 26908943
- [Background] Khan R, Spagnoli V, Tardif JC, L'Allier PL. Novel anti-inflammatory therapies for the treatment of atherosclerosis. Atherosclerosis. 2015 Jun;240(2):497-509. doi: 10.1016/j.atherosclerosis.2015.04.783. Epub 2015 Apr 18. PMID 25917947
- [Background] Prodanovich S, Ma F, Taylor JR, Pezon C, Fasihi T, Kirsner RS. Methotrexate reduces incidence of vascular diseases in veterans with psoriasis or rheumatoid arthritis. J Am Acad Dermatol. 2005 Feb;52(2):262-7. doi: 10.1016/j.jaad.2004.06.017. PMID 15692471
- [Background] Barnabe C, Martin BJ, Ghali WA. Systematic review and meta-analysis: anti-tumor necrosis factor alpha therapy and cardiovascular events in rheumatoid arthritis. Arthritis Care Res (Hoboken). 2011 Apr;63(4):522-9. doi: 10.1002/acr.20371. PMID 20957658
- [Background] Vaidya K, Arnott C, Martinez GJ, Ng B, McCormack S, Sullivan DR, Celermajer DS, Patel S. Colchicine Therapy and Plaque Stabilization in Patients With Acute Coronary Syndrome: A CT Coronary Angiography Study. JACC Cardiovasc Imaging. 2018 Feb;11(2 Pt 2):305-316. doi: 10.1016/j.jcmg.2017.08.013. Epub 2017 Oct 18. PMID 29055633
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Ridker PM, Everett BM, Pradhan A, MacFadyen JG, Solomon DH, Zaharris E, Mam V, Hasan A, Rosenberg Y, Iturriaga E, Gupta M, Tsigoulis M, Verma S, Clearfield M, Libby P, Goldhaber SZ, Seagle R, Ofori C, Saklayen M, Butman S, Singh N, Le May M, Bertrand O, Johnston J, Paynter NP, Glynn RJ; CIRT Investigators. Low-Dose Methotrexate for the Prevention of Atherosclerotic Events. N Engl J Med. 2019 Feb 21;380(8):752-762. doi: 10.1056/NEJMoa1809798. Epub 2018 Nov 10. PMID 30415610
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Moura JA, Valduga CJ, Tavares ER, Kretzer IF, Maria DA, Maranhao RC. Novel formulation of a methotrexate derivative with a lipid nanoemulsion. Int J Nanomedicine. 2011;6:2285-95. doi: 10.2147/IJN.S18039. Epub 2011 Oct 12. PMID 22072866
- [Background] Bulgarelli A, Martins Dias AA, Caramelli B, Maranhao RC. Treatment with methotrexate inhibits atherogenesis in cholesterol-fed rabbits. J Cardiovasc Pharmacol. 2012 Apr;59(4):308-14. doi: 10.1097/FJC.0b013e318241c385. PMID 22113347
- [Background] Hansson GK, Libby P. The immune response in atherosclerosis: a double-edged sword. Nat Rev Immunol. 2006 Jul;6(7):508-19. doi: 10.1038/nri1882. Epub 2006 Jun 16. PMID 16778830
- [Background] Hansson GK. Inflammation and Atherosclerosis: The End of a Controversy. Circulation. 2017 Nov 14;136(20):1875-1877. doi: 10.1161/CIRCULATIONAHA.117.030484. Epub 2017 Sep 15. No abstract available. PMID 28916641
- See also: World Health Organization (WHO) — http://www.who.int/mediacentre/factsheets/fs317/en/